CLINICAL TRIAL: NCT02463149
Title: Pilot Evaluation of Youth Chef Academy: A Plant-based Cooking Program for Urban Middle School Students
Brief Title: Pilot Evaluation of Youth Chef Academy
Acronym: YCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Milwaukee (Other)
Responsible Party: Principal Investigator, Amy Harley, Associate Professor, University of Wisconsin, Milwaukee
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRJ49IH; 11.336 (Other: UW-Milwaukee IRB)
Record Dates: First submitted 2015-06-01; First posted 2015-06-04 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Dietary Modification; Child
Keywords: School health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Youth Chef Academy (Experimental): Receives intervention
  Interventions: Behavioral: Youth Chef Academy
- Control (No Intervention): Usual classroom curriculum

INTERVENTIONS:
Behavioral: Youth Chef Academy — Nutrition and culinary curriculum delivered in the classroom
  Arms: Youth Chef Academy

SUMMARY:
This project examined the effectiveness of Youth Chef Academy (YCA), a classroom-based experiential culinary and nutrition literacy curriculum for middle-school students. The primary study hypothesis was that students assigned to YCA would demonstrate greater improvement in F/V and whole grain consumption compared to students in the control group. Eight classrooms in eight public K-8 schools participated in the project. Classrooms were assigned to intervention or control condition in a non-randomized manner. YCA was delivered by project staff to all of the students in the four intervention classrooms. Students completed a survey to assess primary and secondary outcomes at baseline, six-week curriculum completion, and at twelve-week curriculum completion (YCA extended twelve-week curriculum cohort).

ELIGIBILITY:
Inclusion Criteria:

* Student in intervention or control classroom

Exclusion Criteria:

-

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 248 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change in fruit and vegetable consumption | Baseline, 6 weeks, 12 weeks
  Change in fruit and vegetable consumption calculated from self-reported times per day consuming fruits and vegetables using the 7-item tool from the Youth Risk Behavioral Surveillance System
Change in whole grain consumption | Baseline, 6 weeks, 12 weeks
  Change in whole grain consumption calculated from self-reported times per day consuming whole grains using a revised version of the 8-item tool from the Power of 3 project